CLINICAL TRIAL: NCT07148778
Title: Evaluation of the Effectiveness of a Chatbot-Supported Web-Based Postpartum Care Package Program for Postpartum Women
Brief Title: Effectiveness of Chatbot-Supported Web Program in Postpartum Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emine Ilkin Aydin (Other)
Responsible Party: Sponsor-Investigator, Emine Ilkin Aydin, Lecturer, Bozok University
Organization: Bozok University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17/04/2025-04/1228-AYBU-001
Record Dates: First submitted 2025-08-13; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Postpartum Care; Web-based Training; Chatbot-Based Training
Keywords: postpartum care
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Chatbot-Assisted Web-Based Postpartum Care Package Program (Experimental)
  Interventions: Behavioral: Educational intervention
- Arm 2: Standard Postpartum Care (No Intervention)

INTERVENTIONS:
Behavioral: Educational intervention — In this study, a web-based postpartum care package program supported by a chatbot will be administered to the intervention group.
  A pre-test will be administered to participants in the intervention group within 24-48 hours after birth.
  Participants in this group will be informed that they must watch the videos in the educational modules until the sixth week postpartum. Reminder messages will also be sent to participants via the website, email, and phone calls (between days 7 and 14 postpartum and week 3 postpartum). Participants who have completed the module training will be eligible for post-tests at 6 weeks postpartum and 3 months postpartum.
  Arms: Arm 1: Chatbot-Assisted Web-Based Postpartum Care Package Program

SUMMARY:
The purpose of this clinical study was to evaluate the effectiveness of a web-based "Postpartum Care Package" program developed for postpartum women and delivered via a chatbot, and to examine its effects on the postpartum health of mothers and newborns.

The key questions it aims to answer are:

* What is the impact of the chatbot-supported web-based "Postpartum Care Package" program on the postpartum health of mothers and newborns?
* Does the chatbot-supported web-based "Postpartum Care Package" program increase women's accessibility and availability of postpartum care resources?

ELIGIBILITY:
Inclusion Criteria: Women who will be included in the study.

* Have given birth between the 37th and 41st weeks of pregnancy,
* Be primigravida,
* Have not been diagnosed with a high-risk pregnancy,
* Have an educational level of primary school or above,
* Have no communication difficulties or mental disabilities,
* Have access to equipment (mobile phone, computer, tablet, internet) for web-based education,
* Have experienced no complications in the mother or baby during pregnancy, childbirth, or the postpartum period,
* Voluntarily agree to participate in the study,

Exclusion Criteria:

* Women who moved outside the province where the study was conducted during the implementation period,
* Women who voluntarily withdrew from the study,
* Women who did not participate in any phase of the study will not be included in the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Individuals who are biologically female and in the postpartum period can participate in the study.
Enrollment: 102 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Postpartum Physical Symptom Severity Scale | Pre-test/24-48 hours postpartum Post-test/6 weeks and 3 months postpartum
  Maternal physical health will be assessed using the Postpartum Physical Symptom Severity Scale. This four-point Likert-type scale ranges from 0 to 54, with higher scores indicating greater severity of postpartum physical symptoms.
Visual Analog Scale | Pre-test/24-48 hours postpartum Post-test/6 weeks and 3 months postpartum
  Mothers' physical discomfort/pain levels will be assessed using a Visual Analog Scale. The scale consists of a 10 cm horizontal line, where "0" represents no discomfort and "10" represents the most severe discomfort imaginable. Participants will be asked to mark the point on the line that best reflects their level of physical discomfort/pain during the assessment. Higher scores indicate more severe discomfort/pain.
Edinburgh Postpartum Depression Scale | Pre-test/24-48 hours postpartum Post-test/6 weeks and 3 months postpartum
  The Edinburgh Postnatal Depression Scale will be used to screen for depressive symptoms in postpartum women. The scale consists of 10 items on a four-point Likert-type scale. Each item is scored from 0 to 3, and the total score ranges from 0 to 30. Higher scores indicate more depressive symptoms.
Sexual Life Quality Scale | Pre-test/24-48 hours postpartum Post-test/6 weeks and 3 months postpartum
  The Sexual Quality of Life Scale will be used to evaluate the impact of sexual functions on the quality of life of individuals. It assesses physical, emotional, and relational aspects of sexual well-being. This Likert-type scale consists of 18 items. Higher scores reflect better sexual quality of life, while lower scores indicate deterioration in sexual well-being.
Breastfeeding Self-Efficacy Scale | Pre-test/24-48 hours postpartum Post-test/6 weeks and 3 months postpartum
  The Breastfeeding Self-Efficacy Scale will be used to assess mothers' levels of breastfeeding self-efficacy. It evaluates maternal perceptions regarding their skills, knowledge, and coping abilities related to breastfeeding. The scale consists of 14 items rated on a five-point Likert scale. Scores range from 14 to 70, with higher scores indicating greater breastfeeding self-efficacy.

SECONDARY OUTCOMES:
Postpartum care package program satisfaction | 3rd month postpartum
  Participants' satisfaction level with the Chatbot-supported web-based Postpartum Care Package program will be measured with a 5-point Likert-type satisfaction survey.

CONTACTS AND LOCATIONS:
Overall Officials: Emine ILKIN AYDIN, Lecturer, Principal Investigator — Yozgat Bozok University

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data (IPD). If data sharing becomes possible in the future, it will be done in accordance with ethical principles and participant confidentiality.